CLINICAL TRIAL: NCT00185315
Title: Open-label, Uncontrolled, Long-term Surveillance Study of Iloprost Aerosol Inhalation Therapy in the Treatment of Patients With Primary or Secondary Pulmonary Hypertension. Follow-up Program for Patients Who Completed 12 Weeks in Study ME97218/300180.
Brief Title: Safety Follow-up Study of Inhaled Iloprost in Patients With Pulmonary Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 90570; 303045; Follow-up 90419-300180
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Iloprost

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Ventavis (Iloprost, BAYQ6256)

INTERVENTIONS:
Drug: Ventavis (Iloprost, BAYQ6256) — Inhaled iloprost

SUMMARY:
The aim of this study is to monitor long-term safety and tolerability of iloprost aerosol inhalation therapy in patients suffering from pulmonary hypertension.

DETAILED DESCRIPTION:
This study has previously been posted by Schering AG, Germany. Schering AG has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the 12-week treatment period of the predecessor Schering study 97218/300180
* Investigator judged iloprost aerosol therapy warranted as a suitable treatment for the respective patient
* Negative pregnancy test for females

Exclusion Criteria:

* Any condition during 12-week treatment period of the predecessor Schering study 97218/300180 that prevents participation in the follow-up safety surveillance study

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2000-02; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Adverse events | Throughout the whole study

SECONDARY OUTCOMES:
Tolerability of treatment | Over a minimum of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (16):
- Belgium (2):
  - Brussels
  - Leuven
- France (5):
  - Clamart
  - Grenoble
  - Lille
  - Reims
  - Tours
- Italy (3):
  - Bologna, BO
  - Montescano, Pavia
  - Pisa, PI
- Amsterdam, Netherlands
- Warsaw, Poland
- Portugal (2):
  - Coimbra
  - Vila Nova de Gaia
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid